CLINICAL TRIAL: NCT06341946
Title: Role of Endoscopic Third Ventriculostomy in Management of Malfunctioning Ventriculoperitoneal Shunt
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Omar Mahmoud Abdellah, assistant lecturer, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-02-05MD
Record Dates: First submitted 2024-03-07; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Hydrocephalus; Shunt Malfunction
Keywords: endoscopic third ventriculostomy
MeSH Terms: conditions — Hydrocephalus | interventions — Ventriculostomy

STUDY DESIGN:
Intervention Model Description: All patients with malfunctioning VP shunt will be included in this study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endoscopic third ventriculostomy (Other): endoscopic third ventriculostomy in patients with malfunctioning ventriculoperitoneal shunt
  Interventions: Device: Endoscopic third ventriculostomy

INTERVENTIONS:
Device: Endoscopic third ventriculostomy — role of endoscopic third ventriculostomy in management of malfunctioning ventriculoperitoneal shunt

SUMMARY:
The aim of this study is to analyze our experience in management of malfunctioning ventriculoperitoneal shunt by using endoscopic third ventriculostomy (ETV).

DETAILED DESCRIPTION:
Cerebrospinal fluid shunting remains the most common line of treatment for hydrocephalus. Endoscopic third ventriculostomy (ETV) is an alternative to cerebrospinal fluid (CSF) shunting that is potentially favorable due to the lack of implanted hardware. Most previous studies of ETV have focused on its role as an initial treatment for hydrocephalus and on comparing ETV with CSF shunting. However ,some patients who have previously been treated with a CSF shunt then developed malfunction are candidate for ETV.

The ETV Success Score (ETVSS) is the most widely used scale to estimate the likelihood of ETV success for a given patient .

Although the age of the patient is the most important component of the ETVSS, history of previous treatment with a shunt is also included in the model. According to the ETVSS, previous shunting reduces the likelihood of ETV success by approximately 10%.

There have been numerous previous studies of ETV in patients with a history of a CSF shunt (post shunt ETV), reporting success rates from 50% to 80% . Two review articles also covered this topic, one of which reported ETV success by meta-analysis in 68% of 519 pooled patients .

Most patients with shunt malfunction and or infection are treated with revision procedures, but ETV can be used as an alternative treatment in such cases .The role of endoscopic management of hydrocephalus in shunt malfunction was not investigated extensively so far.

There are several studies which have considered ETV as the main treatment of hydrocephalus inpatients with shunt failure.

Therefore, this is an attractive topic in neurosurgery especially in pediatric neurosurgery that can work and make a different kind of studies to explore the role of ETV for shunt failure.

The goal of the current study was to present our experience with endoscopic third ventriculostomy for management of shunt malfunction.

ELIGIBILITY:
Inclusion Criteria:

* • All patients with malfunctioning VP shunt will be included in this study.

Exclusion Criteria:

* Patients with contraindications for endoscopic procedure such as intracranial infection or bleeding disorders
* Previous unsuccessful attempts of endoscopic third ventriculostomy.
* Active infection or inflammation in the central nervous system.
* Recent history of intracranial hemorrhage.
* Medically unfit for surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-05 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Glasgow Coma Scale (GCS) | base line
  clinical symptoms improvement this Score has values between 3 and 15, 3 being the worst and 15 being the highest
visual analogue scale( VAS ) | base line
  clinical symptoms improvement this Score has values between 0 and 10, 0 being the best and 10 being the worst
visual acuity | base line
  clinical symptoms improvement

SECONDARY OUTCOMES:
radiological CT brain and or MRI brain | base line
  CT brain and or MRI brain

REFERENCES:
- [Background] Kulkarni AV, Drake JM, Kestle JR, Mallucci CL, Sgouros S, Constantini S; Canadian Pediatric Neurosurgery Study Group. Predicting who will benefit from endoscopic third ventriculostomy compared with shunt insertion in childhood hydrocephalus using the ETV Success Score. J Neurosurg Pediatr. 2010 Oct;6(4):310-5. doi: 10.3171/2010.8.PEDS103. PMID 20887100
- [Background] Kulkarni AV, Riva-Cambrin J, Browd SR. Use of the ETV Success Score to explain the variation in reported endoscopic third ventriculostomy success rates among published case series of childhood hydrocephalus. J Neurosurg Pediatr. 2011 Feb;7(2):143-6. doi: 10.3171/2010.11.PEDS10296. PMID 21284458
- [Background] Furtado LMF, da Costa Val Filho JA, Holliday JB, da Silva Costa J, de Matos MA, Nascimento VAM, Ramos Cavalcanti T. Endoscopic third ventriculostomy in patients with myelomeningocele after shunt failure. Childs Nerv Syst. 2020 Dec;36(12):3047-3052. doi: 10.1007/s00381-020-04596-5. Epub 2020 Apr 4. PMID 32248278
- [Background] Takeshige N, Uchikado H, Nakashima D, Negoto T, Nagase S, Yoshitomi M, Sakata K, Morioka M. Endoscopic third ventriculostomy for myelomeningocele-related hydrocephalus after shunt failure: Long-term outcome in a series of 8 patients. Clin Neurol Neurosurg. 2021 Feb;201:106406. doi: 10.1016/j.clineuro.2020.106406. Epub 2020 Dec 4. PMID 33341457
- [Background] Chhun V, Sacko O, Boetto S, Roux FE. Third Ventriculocisternostomy for Shunt Failure. World Neurosurg. 2015 Jun;83(6):970-5. doi: 10.1016/j.wneu.2015.01.058. Epub 2015 Mar 13. PMID 25772610
- [Background] Irrinki RNNS, Bawa M, Hegde S, Chhabra R, Gupta V, Gupta SK. Functional and Radiological Parameters to Assess Outcome of Endoscopic Third Ventriculostomy in Shunt Failure Patients. J Pediatr Neurosci. 2019 Apr-Jun;14(2):65-69. doi: 10.4103/jpn.JPN_31_19. PMID 31516622
- [Background] Talamonti G, Nichelatti M, Picano M, Marcati E, D'Aliberti G, Cenzato M. Endoscopic Third Ventriculostomy in Cases of Ventriculoperitoneal Shunt Malfunction: Does Shunt Duration Play a Role? World Neurosurg. 2019 Jul;127:e799-e808. doi: 10.1016/j.wneu.2019.03.268. Epub 2019 Apr 4. PMID 30954740
- [Background] Boschert J, Hellwig D, Krauss JK. Endoscopic third ventriculostomy for shunt dysfunction in occlusive hydrocephalus: long-term follow up and review. J Neurosurg. 2003 May;98(5):1032-9. doi: 10.3171/jns.2003.98.5.1032. PMID 12744363
- [Background] Bilginer B, Oguz KK, Akalan N. Endoscopic third ventriculostomy for malfunction in previously shunted infants. Childs Nerv Syst. 2009 Jun;25(6):683-8. doi: 10.1007/s00381-008-0779-1. Epub 2008 Dec 11. PMID 19082608